CLINICAL TRIAL: NCT05629832
Title: Transpulmonary Pressure Guided Mechanical Ventilation Strategy for Right Ventricle Protection in Acute Respiratory Distress Syndrome
Brief Title: Transpulmonary Pressure in Right Ventricle Protection of ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Xiao Tang, Doctor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ptp right ventricle protection
Record Dates: First submitted 2022-11-14; First posted 2022-11-29 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Cor Pulmonale
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTP group (Experimental)
  Interventions: Procedure: mechanical ventilation strategy guided by transpulmonary pressure
- Control group (No Intervention)

INTERVENTIONS:
Procedure: mechanical ventilation strategy guided by transpulmonary pressure — Mechanical ventilation parameters adjust guided by transpulmonary pressure monitoring. For pressure assist control or volumn assit control mode; inspiratory pressure or volumn setting needs to maintain Ppeak less than 25 cm H2O; PEEP was set at such a level that expiratory Ptp stayed between 0 and 5 cm H2O.
  Arms: PTP group

SUMMARY:
To compare the effect between mechanical ventilation strategy guided by transpulmonary pressure and tranditional lung protective ventilation strategy in acute respiratory distress syndrome for right ventricle protection.

ELIGIBILITY:
Inclusion Criteria:

* duration of invasive mechanical ventilation less than 72 hours;
* meet the diagnostic criteria of Berlin definition for ARDS;
* age older than 18

Exclusion Criteria:

* esophageal surgery or damage;
* cardiac surgery;
* severe bronchopleural fistula;
* serious arrhythmia; pneumothorax;
* tricuspid stenosis;
* heparin allergy;
* chronic pulmonary heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular resistance (PVR) | 3 days
  PVR will measured by Swan-Ganz catheter
Pulmonary vascular compliance | 3 days
  Pulmonary vascular compliance will be calculated using pulmonary artery pressure divided by stroke output measured by Swan-Ganz catheter.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided